CLINICAL TRIAL: NCT01434082
Title: Sleep Patterns in Children With and Without Juvenile Idiopathic Arthritis
Acronym: JIA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Teresa Ward, Assistant Professor, Prinicpal Investigator, University of Washington
Other Study IDs: JIA; 1R01NR012734-01 (NIH)
Record Dates: First submitted 2011-09-09; First posted 2011-09-14 (Estimated); Last update posted 2011-09-14 (Estimated); Status verified 2011-09

CONDITIONS: Juvenile Idiopathic Arthritis
Keywords: sleep; school-age children; Children with and without arthritis
MeSH Terms: conditions — Arthritis, Juvenile

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Morning urine and saliva
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: comparison of types of sleep disordered breathing — comparison of types of sleep disordered breathing (primary snoring, upper airway resistance syndrome, obstructive sleep apnea) in children with and without arthritis.

SUMMARY:
The investigators are doing this study to look at sleep problems, daytime sleepiness, and thinking and behavior patterns in children with arthritis and in children without arthritis. Arthritis is a problem with joints. Some children have arthritis and some children do not have arthritis.

Sleep disordered breathing is a sleeping problem in which some children snore and have pauses in their breathing during sleep. It is associated with not enough or fragmented sleep, poor school performance, problems paying attention, and behavior problems.

The investigators do not know how many children with arthritis have sleep problems, and how it is linked to daytime sleepiness and children's learning, and behavior patterns compared to children without arthritis. The investigators need to study both children with arthritis and children without arthritis to learn more about these connections and to understand if they are the same or different in children with arthritis and in children without arthritis.

DETAILED DESCRIPTION:
Overview of Study:

* Children and their parent will be scheduled to come to the University of Washington School of Nursing Sleep Laboratory for overnight polysomnography, and to complete multi-sleep latency tests and a battery of neurobehavioral performance tests the next day at a convenient time and day.
* Children will be asked to complete a sleep, symptoms (pain, fatigue), behavior, and day to day activity surveys, and the parent who accompanies the child to the laboratory, will be asked to complete surveys assessing demographics, child's usual sleep, behavior, school performance, health status, and family functioning.
* Children will also be asked to spit in a container and urinate in a container upon awakening in the morning after their sleep study.

Primary Aims of the Study:

1. Compare indices of sleep disturbances, risk factors, and type of sleep disordered breathing(primary snoring, upper airway resistance syndrome, obstructive sleep apnea) in Juvenile Idiopathic Arthritis (JIA) to age, sex matched control children.
2. Compare scores on neurobehavioral tests and daytime sleepiness; and to describe associations between indices of sleep disturbances on neurobehavioral performance and daytime sleepiness in JIA to age, sex matched control children.

Secondary Objectives:

1. Describe and compare parent report of child's sleep habits, fatigue, behavior, school performance, day-to-day activity, and family functioning in children with JIA to age, sex matched control children.

ELIGIBILITY:
Inclusion Criteria:

Children

* Children with and without arthritis, 6 thru 11 years old, able to speak English
* Children with JIA not recently hospitalized for severe JIA.

Parents

* Subject's parents or legal guardian are > 18 years of age and able to read and speak English.
* Subject's parent or legal guardian has provided written informed consent prior to screening for this study.

Exclusion Criteria:

Children

* A child with a history of/current diagnosis of a psychiatric condition meeting DSM-IV-TR (e.g. depression, bipolar disorder) that would interfere with ability to comply with protocol requirements, or give informed consent, or be expected to have disordered sleep.
* A child with acute illness such as a cold or the flu that would interfere with sleep and neurobehavioral testing.
* A chronic condition such as cancer, diabetes, or asthma which would, in the investigator's opinion, compromise the subject's ability to comply with the study requirements and interfere with ability to comply with protocol requirements.
* Children admitted to the hospital for severe JIA within the last 2 months.
* Children with a BMI >95th percentile (defined as obesity by CDC) will be excluded because of potential impact of obesity on SDB.

Parents

* A parent or legal guardian with a chronic condition that would compromise the parent's ability to comply with protocol requirements.

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: * Children with arthritis will be recruited from the Division of Pediatric Rheumatology at Seattle Children's Hospital.
  * Children without arthritis will be recruited from the King COunty community.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2011-09; Primary Completion 2015-01 (Estimated); Study Completion 2015-02 (Estimated)

PRIMARY OUTCOMES:
Prevalence of Sleep Disordered Breathing | 3.5 years

SECONDARY OUTCOMES:
Measures of Daytime Sleepiness | 3.5 years
  After the overnight sleep study, children will undergo multiple sleep latency tests which are four 20-minute nap opportunities that assess daytime sleepiness.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Washington School of Nursing, Seattle, Washington, United States